CLINICAL TRIAL: NCT03687424
Title: The Effect of High-flow Nasal Oxygenation vs. Low-flow Nasal Oxygenation on Oxygen Saturation During Analgo-sedation in Obese Adult Patients, Randomized Controlled Trial
Brief Title: Can High-flow Nasal Oxygenation Improve Oxygen Saturation During Analgo-sedation in Obese Adults?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Split, School of Medicine (Other)
Collaborators: General Hospital Dubrovnik (Other)
Responsible Party: Principal Investigator, Anita Vukovic, MD, specialist of anesthesiology, reanimatology and intensive care, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-285/8-3-17-B
Record Dates: First submitted 2018-09-22; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Noninvasive Ventilation; Respiratory Insufficiency; Obesity; Deep Sedation; Hypoxia; Airway Management; Colonoscopy
Keywords: "Noninvasive Ventilation"[Mesh]; "Obesity"[Mesh]; "Deep Sedation"[Mesh]; "Hypoxia"[Mesh]; "Adult"[Mesh]; "Airway management"[Mesh]; "Colonoscopy"[Mesh]
MeSH Terms: conditions — Respiratory Insufficiency; Obesity; Hypoxia

STUDY DESIGN:
Intervention Model Description: We plan to conduct prospective, parallel group, randomized controlled clinical trial.
  In total, 126 participants will be included in this trial. These participants are patients scheduled for outpatient colonoscopy in analgo-sedation.
  This study includes 126 patients divided in 3 groups of according to BMI: 18<BMI<30 kg/m2, 30<BMI<40 kg/m2 or BMI ≥40 kg/m2. Each group will be divided in control groups of 21 patients who will receive LFNO and intervention groups of 21 patients who will receive HFNO during standardized intravenous analgo-sedation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Anesthesiologist who interviews and examines patients scheduled for colonoscopy under analgo-sedation will enroll eligible participants and will offer procedure explanation and possibility to sign uniformed written consent. Unique personal hospital admission number (UPHAN) will be assigned to all eligible participants. After that, they will be randomized to control or intervention group by using random numbers generator. Anesthesiologist who implements anesthesia will receive nontransparent envelope with assigned intervention provided by independent investigator and will not decide which participant will receive LFNO or HFNO. However, attending anesthesiologist and participants will unavoidably be aware of type of oxygenation applied. Investigator who collects data after procedure will be unaware of study protocol and will enter data to formatted database. Participants' data will be noted under UPHAN. Outcome assessors will be unaware of intervention applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Normal weight 18<BMI<30 kg/m2 LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- Obese 30<BMI<40 kg/m2 LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- Morbidly obese BMI ≥40 kg/m2 LFNO (Active Comparator): Low-flow nasal oxygenation (LFNO) O2 flow 5L/min, FiO2 40%
  Interventions: Device: low-flow nasal oxygenation (LFNO)
- Normal weight 18<BMI<30 kg/m2 HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)
- Obese 30<BMI<40 kg/m2 HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)
- Morbidly obese BMI ≥40 kg/m2 HFNO (Experimental): High-flow nasal oxygenation (HFNO) O2 flow 40L/min, FiO2 40%
  Interventions: Device: high-flow nasal oxygenation (HFNO)

INTERVENTIONS:
Device: high-flow nasal oxygenation (HFNO) — Experimental HFNO: O2 flow 40L/min, FiO2 40%
  Arms: Morbidly obese BMI ≥40 kg/m2 HFNO; Normal weight 18<BMI<30 kg/m2 HFNO; Obese 30<BMI<40 kg/m2 HFNO
Device: low-flow nasal oxygenation (LFNO) — Active comparator (LFNO): O2 flow 5L/min, FiO2 40%
  Arms: Morbidly obese BMI ≥40 kg/m2 LFNO; Normal weight 18<BMI<30 kg/m2 LFNO; Obese 30<BMI<40 kg/m2 LFNO

SUMMARY:
Obesity is omnipresent problem in everyday anesthesiology practice associated with low level of blood oxygen (hypoxemia) during analgo-sedation. Overweight outpatients are often scheduled for colonoscopy usually undergo analgo-sedation. In obese patients, intravenous analgo-sedation often diminish respiratory drive causing hypoxemia. To avoid hypoxemia, low-flow nasal oxygenation (LFNO) of 2-6 L/min is applied via standard nasal catheter to provide maximum 40 % of inspired fraction of oxygen (FiO2). LFNO comprises applying cold and dry oxygen which causes discomfort to nasal mucosa of patient. LFNO is often insufficient to provide satisfying oxygenation. Insufficient oxygenation adds to circulatory instability - heart rate (HR) and blood pressure (BP) disorder.

On the other side, high-flow nasal oxygenation (HFNO) brings 20 to 70 L/min of heated and humidified of O2/air mixture up to 100% FiO2 via specially designed nasal cannula. Heated and humidified O2/air mixture is much more agreeable to patient. HFNO brings noninvasive support to patients' spontaneous breathing by producing continuous positive pressure of 3-7 cmH2O in upper airways consequently enhancing oxygenation.

Investigators intend to analyze effect of HFNO vs. LFNO on oxygen saturation during procedural analgo-sedation for colonoscopy in obese adult patients.

Investigators expect that obese patients with preserved spontaneous breathing, oxygenized by HFNO vs. LFNO, will be less prone to hypoxemia thus more respiratory and circulatory stable during procedural analgo-sedation for colonoscopy.

Obese patients with applied HFNO should longer preserve: normal oxygen saturation, normal level of CO2 and O2, reflecting better respiratory stability. Investigators expect obese participnts to have more stable HR and BP, reflecting improved circulatory stability. There will be less interruption of breathing pattern of obese patients and less necessity for attending anesthesiologist to intervene.

DETAILED DESCRIPTION:
Obese patients are often scheduled for colonoscopy under analgo-sedation. Analgo-sedation is characterized by deep conscious sedation and preserved spontaneous breathing. Continuous intravenous application of sedatives favors patients' circulatory stability and application of oxygenation contributes to maintaining adequate patients' oxygenation. Typically, low-flow nasal oxygenation (LFNO) of 2-6 L/min is applied via standard nasal catheter to provide maximum 40% of inspired fraction of oxygen (FiO2) before (preoxygenation), during (procedural oxygenation) and after (postprocedural oxygenation) until patient regains consciousness.

During analgo-sedation obese patients are prone to intervals of bradypnea and hypoventilation. Transitory apnea in obese patients could lead to hypoxemia, hypoxia, hypercapnia and hemodynamic insufficiency despite LFNO application. Fatal outcome may occur, especially at higher risk overweight patients (ASA III class). Respiratory and hemodynamic stability of morbidly obese outpatients during analgo-sedation for endoscopic procedures represent challenge to anesthesiologists. There is no generally accepted protocol of preoxygenation and intraoperative ventilatory management for obese patients. Obese (30<BMI<40 kg/m2, BMI= body mass index) and morbidly obese patients (BMI ≥40 kg/m2) are classified to higher anesthesia risk groups, even if obese patients may not have other comorbidities (30<BMI<40 kg/m2 = ASA II, BMI ≥40 kg/m2 = ASA III).

Partial relaxation of pharyngeal muscles characteristic for analgo-sedation in overweight patients causes prolapse of fatty tissue that partially obstructs pharynx and can cause obstructive sleep apnoea (OSA). Although OSA is not related to obesity, OSA can accompany obesity. Besides perioperatively, hypoxia and bradypnoea episodes occur postoperatively in obese patients, which makes additional observation of obese patients necessary. More frequent hypoxia and bradypnoea during awakening require additional respiratory effort. Ventilation strategies in obese patients are necessary to optimize gas exchange and pulmonary mechanics in order to reduce pulmonary complications.

High-flow nasal oxygenation (HFNO) brings 20 to 70 L/min heated and humidified O2/air mixture up to 100% FiO2 via specially designed, soft nasal cannula. HFNO brings non-invasive support to patients' inspiratory effort by developing 3-7 cmH2O of continuous pressure in upper airway, decreasing it's resistance and dead space. Also, heated and humidified oxygen/air mixture with possibility to bring higher FiO2 adds to better patients' oxygenation preservation and improved patients' comfort during procedure.

AIM of this study is to compare effect of HFNO vs. LFNO during standardized procedure of intravenous analgo-sedation on periprocedural oxygenation maintenance in patients of different weight groups: 18<BMI<30 kg/m2, 30<BMI<40 kg/m2 and BMI ≥40 kg/m2.

Investigators hypothesized that application of HFNO compared to LFNO, in obese patients with preserved spontaneous breathing during procedural analgo-sedation, contributes to maintaining adequate oxygenation, consequently adding to greater peri-procedural circulatory and respiratory stability of obese patients. Investigators expect that HFNO will ensure reduced bradypnoea intervals (frequency of breathing, FoB 1/min), longer maintenance of adequate oxygenation, shorter intervals of desaturation (SpO2 ≤ 92%), reducing hypercapnia (PaCO2 ≥ 6 kPa) and less airway - opening maneuvers performed by attending anesthesiologist (Aom). These will prevent partial respiratory insufficiency detected by low SpO2 or low PaO2 ≤ 11 kPa accompanied by normal or low PaCO2 ≤ 6 kPa, and global respiratory insufficiency detected by decreased SpO2 ≤ 92% and PaO2 ≤ 11 kPa with increased PaCO2 ≥ 6 kPa.

Investigators plan to conduct prospective, parallel group, randomized controlled clinical trial. Trial will be managed according to principles of Declaration of Helsinki for scientific clinical research and will be planned and guided according to CONSORT guidelines (Consolidated Standards of Reporting Trials). The trial has been approved by hospital's Ethic Committee.

The source of information are going to be 126 adult patients scheduled for colonoscopy under analgo-sedation in the setting of daily outpatient gastroenterology ambulance. Eligible participants will be interviewed and examined ambulatory by anesthesiologist together with evaluation of ASA status, difficulty of airway management and BMI. After initial examination inclusive and exclusive criteria will be distinguished. Eligible participants who give written consent of participation will be included in this trial. After that, participants will be assigned to equal normal weight (18<BMI<30 kg/m2), obese (30<BMI<40 kg/m2) or morbidly obese (BMI ≥40 kg/m2) group. Each group will be randomized to intervention (HFNO) and control (LFNO) subgroup by random numbers generator. Randomization will be used until adequate number of participants in every group is reached.

Interventions: intervention subgroups participants will be oxygenated via nasal cannula using high flow (40 L/min) of humidified and heated oxygen in air mixture (FiO2 40%). HFNO will be applied by oxygenator (AirVO™2, Fisher and Paykell, New Zealand, Technomedika Croatia d.o.o.) during procedural analgo-sedation for colonoscopy with maintained spontaneous breathing. In control subgroups, oxygenation will be applied via nasal catheter (Bauerfeind d.o.o, Zagreb, Croatia) using standard low flow oxygen (5 L/min, FiO2 40%) LFNO. In both groups concentration of oxygen delivered depends on oxygen flow which is regulated by standard flow-regulator (flowmeter). Oxygen is delivered through pipelines from central hospital gas supply or from portable cylinder gas supply.

Anesthesia procedure will be uniformed for all participants. Integrated noninvasive monitoring of vital functions will be set: EKG - (heart rate/min), SpO2 (%), blood pressure (mmHg), indirect respiration (number of breaths/min) (Compact 7; Medical Econet GmbH, Germany).

Every participant will have established intravenous infusion of 250 ml NaCl 0.9% through intravenous cannula regulated by continuous flow (Extension set/CONTROL-A-FLO Regulator 19" Male Luer Lock Adapter, Baxter/Agmar d.o.o. United States of America/Croatia).

Arterial cannula (REF30401, 20 G - 1,10 mm x 45 mm 49 ml, atraumatic needle tip, Medbar LTD, Izmir, Turkey) will be placed in radial artery in a previously anesthetized area with local anesthetic (EMLA).

Oxygenation (HFNO or LFNO) will be administrated in continuity until patients' awakening. Oxygenation will be started 3 minutes before starting analgo-sedation (preoxygenation), continued during analgo-sedation and procedure of colonoscopy (perioperative oxygenation) and up to five minutes after colonoscopy and until patient is awaken (postprocedural oxygenation).

Intravenous analgo-sedation will be started through continuous infusions of propofol and fentanyl. Induction of sedation will be guided by TCI (Target control Infusion) (B. Braun Melsungen, Germany) with initial target propofol concentration of 6 micrograms/minute. Expected time of induction with this concentration is 60-120 seconds. This target concentration allows hemodynamic and respiratory stability. Required analgesia will be simultaneously applied through slow continuous infusion in dose of 0.05 mcg/kg/min in order to preserve spontaneous breathing. Slow infusion will be applied through perfusor (B.Braun, Melsungen, Germany). Analgo-sedation will be discontinued immediately after end of the procedure.

Control of nasopharyngeal airway passage during procedure is achieved by using oropharyngeal airway, if necessary. Oropharyngeal airway (Airway; Vigon-Medicpro d.o.o.) will be inserted after achieving moderate sedation, and only if base of tongue is closing airway by dropping on posterior pharyngeal wall. Every manipulation of patients' airway by anesthesiologist will be documented (insertion of airway, jaw thrust maneuver).

Sampling: one milliliter of arterial blood will be collected as three consecutive samples from arterial cannula before, during and after analgo-sedation. Sample of arterial blood will be drawn from left radial or cubital artery.

Measurements: measurement of oxygenation will be done using two methods: indirect (noninvasive) method using pulse oxymeter (Compact 7, Medical ECONET GmbH, Germany) and direct (invasive) method from obtained arterial blood sample. Measurement of SpO2 and drawing arterial blood sample will be done simultaneously. Direct measurements of SpO2 and PaO2 will be taken in intervals of time. SpO2 will be measured on the left-hand index finger. Data will be uniformly collected through indirect - noninvasive (SpO2, heart rate, blood pressure, respiratory rate) and direct - invasive (arterial blood gas analysis - pH, PaO2, PaCO2, SaO2) measurements.

Possible biases and confounding variables could be caused by hypothermia of participant, by sphygmomanometer cuff pressure on the same arm where blood samples are drawn and by prolonged time of arterial blood analysis. These difficulties can be bypassed by: adjustment of room temperature where analgo-sedation is performed, blood pressure measuring on opposite arm from where samples of blood are taken and by arterial blood gas analysis without delay.

Basic data analyses will be performed by statistician. Sample size is determined by statistic computing web program: http://www.stat.ubc.ca/~rollin/stats/ssize used statistic test Inference for Proportions: Comparing Two Independent Samples. Assessment of sample size is computed for two independent samples with assumption of clinically significant difference in patients' oxygenation: ≤11 and ≥14.4 kPa with delta 4.4. Statistical significance of difference will be inferred with 5% α-error, 50% β-error and study power 0.80. Calculated size of sample is: 21 participant pro subgroup (total of 126 participants).

Investigators expect no changes to methods after trial commencement. All potential unwanted events which may happen during analgo-sedation and colonoscopy that could cause deviation from this trial's protocol will be reason for exclusion of participant from this trial. If circumstances change, anesthesiologist responsible for application of anesthesia will carry out procedure in way which is in patients' best interest.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (18<BMI<30 kg/m2)
* obese patients (30<BMI<40 kg/m2)
* morbidly obese patients (BMI≥40 kg/m2)
* intravenous analgo-sedation
* elective colonoscopy
* colorectal tumors.

Exclusion Criteria:

* emergency colonoscopy
* diseases of peripheral blood vessels
* hematological diseases
* psychiatric diseases
* sideropenic anemia
* patients' refusal
* ongoing chemotherapy or irradiation
* propofol allergies
* fentanyl allergies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of peripheral blood oxygenation (SpO2), | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Peripheral blood saturation (SpO2):
  Normal range ≥ 92% Acceptable deflection from normal values of peripheral blood saturation (SpO2) significant for hypoxemia is < 92%, while all values above will be considered normal.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of arterial blood saturation (PaO2) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Partial pressure of oxygen (PaO2):
  Normal range: ≥11 kPa Partial pressure of oxygen (PaO2), ≥ 11 kPa PaO2 will be considered normal, while all values below are considered significant for hypoxemia.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.

SECONDARY OUTCOMES:
Change of pH (pH) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  pH value of arterial blood sample :
  Normal values: 7.35 - 7.45. Acceptable deflection from normal values significant for acidosis: pH <7.35.
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of partial pressure of CO2 (PaCO2) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Partial pressure of CO2 (PaCO2):
  Normal range: 4.7 - 6.4 kPa. Acceptable deflection from normal values significant for hypercapnia: PaCO2 ≥ 6 kPa
  Above-mentioned parameter will be observed during procedure so that we can confirm or exclude differences connected with practical application of LFNO and HFNO.
Change of normopnea (FoB) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of breathing. (FoB/min - number of breaths per minute). Normal range: 12 - 20 breaths per minute. Bradypnoea will be noted when number of breaths is less than 12 breaths/min.
Change of frequency of desaturation (fDE) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of desaturation during time of analgo-sedation: (fDE/min, SpO2<92%). Normal range: fDE ≤1/30, up to one episode of desaturation from the start to the end of analgo-sedation. Acceptable deflection from normal range: more than one desaturation in 30 minutes.
Change of duration of desaturation (DE/min) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Duration of desaturation (DE/min). Normal range: up to one minute. Duration of desaturation longer then one minute will be considered as insufficient ventilation.
Change of frequency of bradypnoea during analgo-sedation (fBRP/min) | From the beginning of oxygenation and analgo-sedation till the end of analgo-sedation and oxygenation - complete procedure duration estimated: 35 minutes
  Frequency of bradypnoea during analgo-sedation (fBRP/min), Normal range: fBRP ≤1/30, up to one episode of bradypnoea from the start to the end of analgo-sedation. Acceptable deflection from normal range: > one episode of bradypnoea during 30 minutes.
Change of heart rate (HR/min) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Heart rate (HR/min): normal range 60 -100/min. Acceptable deflection from normal values is < 60 heartbeats/min significant for bradycardia, while all values up to 100 heartbeats per minute will be considered normal.
Change of mean arterial pressure (MAP) | Before procedure: 1 minute before start of analgo-sedation and oxygenation, During procedure: 15 minutes from beginning of oxygenation and analgo-sedation, After procedure: 5 minutes after discontinuing oxygenation and analgo-sedation
  Mean arterial pressure (MAP): normal range: 65 -110 mmHg Acceptable deflection from normal values is < 65 mmHg - significant for hypotension.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becker DE, Haas DA. Management of complications during moderate and deep sedation: respiratory and cardiovascular considerations. Anesth Prog. 2007 Summer;54(2):59-68; quiz 69. doi: 10.2344/0003-3006(2007)54[59:MOCDMA]2.0.CO;2. PMID 17579505
- [Background] Anand GW, Heuss LT. Feasibility of breath monitoring in patients undergoing elective colonoscopy under propofol sedation: A single-center pilot study. World J Gastrointest Endosc. 2014 Mar 16;6(3):82-7. doi: 10.4253/wjge.v6.i3.82. PMID 24634712
- [Background] Lee CC, Perez O, Farooqi FI, Akella T, Shaharyar S, Elizee M. Use of high-flow nasal cannula in obese patients receiving colonoscopy under intravenous propofol sedation: A case series. Respir Med Case Rep. 2018 Feb 3;23:118-121. doi: 10.1016/j.rmcr.2018.01.009. eCollection 2018. PMID 29719796
- [Background] Frieling T, Heise J, Kreysel C, Kuhlen R, Schepke M. Sedation-associated complications in endoscopy--prospective multicentre survey of 191142 patients. Z Gastroenterol. 2013 Jun;51(6):568-72. doi: 10.1055/s-0032-1330441. Epub 2013 Jun 5. PMID 23740356
- [Background] Frat JP, Goudet V, Girault C. [High flow, humidified-reheated oxygen therapy: a new oxygenation technique for adults]. Rev Mal Respir. 2013 Oct;30(8):627-43. doi: 10.1016/j.rmr.2013.04.016. Epub 2013 May 29. French. PMID 24182650
- [Background] Nagata K, Morimoto T, Fujimoto D, Otoshi T, Nakagawa A, Otsuka K, Seo R, Atsumi T, Tomii K. Efficacy of High-Flow Nasal Cannula Therapy in Acute Hypoxemic Respiratory Failure: Decreased Use of Mechanical Ventilation. Respir Care. 2015 Oct;60(10):1390-6. doi: 10.4187/respcare.04026. Epub 2015 Jun 23. PMID 26106206
- [Background] Ni YN, Luo J, Yu H, Liu D, Ni Z, Cheng J, Liang BM, Liang ZA. Can High-flow Nasal Cannula Reduce the Rate of Endotracheal Intubation in Adult Patients With Acute Respiratory Failure Compared With Conventional Oxygen Therapy and Noninvasive Positive Pressure Ventilation?: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):764-775. doi: 10.1016/j.chest.2017.01.004. Epub 2017 Jan 13. PMID 28089816
- [Background] Nathanson V. Revising the Declaration of Helsinki. BMJ. 2013 May 8;346:f2837. doi: 10.1136/bmj.f2837. No abstract available. PMID 23657182
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Background] Groves N, Tobin A. High flow nasal oxygen generates positive airway pressure in adult volunteers. Aust Crit Care. 2007 Nov;20(4):126-31. doi: 10.1016/j.aucc.2007.08.001. Epub 2007 Oct 10. PMID 17931878
- [Background] Gotera C, Diaz Lobato S, Pinto T, Winck JC. Clinical evidence on high flow oxygen therapy and active humidification in adults. Rev Port Pneumol. 2013 Sep-Oct;19(5):217-27. doi: 10.1016/j.rppneu.2013.03.005. Epub 2013 Jul 8. PMID 23845744
- [Background] Jirapinyo P, Thompson CC. Sedation Challenges: Obesity and Sleep Apnea. Gastrointest Endosc Clin N Am. 2016 Jul;26(3):527-37. doi: 10.1016/j.giec.2016.03.001. PMID 27372775
- [Background] Bignami E, Saglietti F, Girombelli A, Briolini A, Bove T, Vetrugno L. Preoxygenation during induction of anesthesia in non-critically ill patients: A systematic review. J Clin Anesth. 2019 Feb;52:85-90. doi: 10.1016/j.jclinane.2018.09.008. Epub 2018 Sep 15. PMID 30227319
- [Background] Shah U, Wong J, Wong DT, Chung F. Preoxygenation and intraoperative ventilation strategies in obese patients: a comprehensive review. Curr Opin Anaesthesiol. 2016 Feb;29(1):109-18. doi: 10.1097/ACO.0000000000000267. PMID 26545146
- See also: American Society of Anesthesiologists (ASA). ASA physical status classification system 2014 Oct [internet]. Schaumburg, Illinois, USA: ASA;2014. — https://www.asahq.org/resources/clinical-information/asa-physical-status-classification-system
- See also: Programiz [internet].Kupandole, Nepal: Parewa Labs Pvt. Ltd. [cited 2018 Sept17]. Flowchart in programming. Available from: — http://www.programiz.com/article/flowchart-programming